CLINICAL TRIAL: NCT05560061
Title: An Uneven Terrain Surface to Improve Locomotor Robustness in People With Amputation
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Substantial redesign of protocol and training warranted new study.
Sponsor: University of Nevada, Las Vegas (Other)
Responsible Party: Principal Investigator, Jenny Kent, Assistant Professor, University of Nevada, Las Vegas
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: UNLV-2021-52
Record Dates: First submitted 2022-09-16; First posted 2022-09-29 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Amputation
Keywords: locomotion; gait; rehabilitation; motor learning; lower limb amputation

STUDY DESIGN:
Intervention Model Description: Participants will be randomized into two groups - 1) uneven - flat; 2) flat - uneven. Uneven and flat sessions will occur on separate days, 12-72 hours apart.
Who Masked: Outcomes Assessor
Masking Description: Outcomes assessor will be blinded to arm.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Uneven terrain walking training (Experimental): Participants will complete walking practice on an uneven terrain surface.
  Interventions: Other: Gait practice on an uneven terrain surface
- Flat terrain walking (Active Comparator): Participants will complete walking practice on a level surface.
  Interventions: Other: Gait practice on a flat terrain surface

INTERVENTIONS:
Other: Gait practice on an uneven terrain surface — Participants will walk back and forth on an uneven terrain surface wearing an overhead harness (with zero bodyweight support), at their self-selected comfortable speed.
  Arms: Uneven terrain walking training
Other: Gait practice on a flat terrain surface — Participants will walk back and forth on a level surface wearing an overhead harness (with zero bodyweight support), at their self-selected comfortable speed.
  Arms: Flat terrain walking

SUMMARY:
To attain high levels of mobility, people with lower limb amputation must build both the skill and the confidence to rely on their prosthesis in the environments that they will encounter in daily life. The purpose of this research is to determine whether practicing walking on an uneven terrain surface, specifically designed to present a modest, manageable disturbance to walking, can improve balance, locomotor flexibility (i.e. the ability to adapt walking to different walking contexts) and balance confidence, to a greater extent than walking on level ground alone. This preliminary study aims to determine whether uneven terrain walking is feasible and acceptable in the target population, and also to establish preliminary efficacy.

DETAILED DESCRIPTION:
The long-term focus of this research is to investigate an uneven terrain training paradigm as an intervention to improve locomotor skill and confidence in lower limb prosthesis users; specifically to determine whether by inducing step-to-step variability in a safe environment, through training on an uneven terrain surface, individuals may develop more adaptable gait, and greater confidence in their mobility. We hypothesize that inducing a manageable level of variability into walking patterns during training will lead to greater balance, locomotor flexibility, and balance confidence. The surface has shallow contours that alter foot-ground interactions at each step, disrupting habitual movement patterns.

The aim of this study is to establish feasibility, acceptability and preliminary efficacy of the uneven surface as a mobility training tool for lower limb prosthesis users. Ambulatory lower limb prosthesis users will attend a biomechanics laboratory on two occasions, during which they will complete walking practice sessions on a flat surface and on an uneven surface. A crossover design will be employed, with walking surface order randomized across participants. Preliminary efficacy will be established based on functional tasks and self-efficacy questions administered before and after the sessions on each day. Feasibility and acceptability will be established based on feasibility study objectives from Orsmond & Cohn's feasibility framework.

ELIGIBILITY:
Inclusion Criteria:

* lower limb amputation at ankle level or above
* properly fitted with a walking prosthesis, used regularly for home and/or community ambulation
* good socket fit assessed by a score of 7-10 on the socket fit comfort score (Hanspal et at., 2003).
* able to walk for two minutes at a time with or without an assistive device
* willing to travel to the test site two times for training and testing.

Exclusion Criteria:

* leg/foot ulcer/sore or other conditions that cause pain during weight-bearing
* cardiovascular, respiratory or other critical health conditions that preclude moderate physical activity
* unilateral or bilateral upper limb absence or loss at the wrist and above
* diagnosis of cognitive disturbances
* allergy to medical adhesives
* women who are pregnant or think they may be pregnant
* acute illness
* dizziness on the day of testing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2025-08-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in single limb stand time from baseline | Pre- and immediately post- training session on day 1 and pre- and immediately post- training session on day 2.
  The duration the participant is able to stand on one limb without touching the floor with the raised foot, out of a maximum of 30 seconds.
Change in balance self-efficacy from baseline | Pre- and immediately post- training session on day 1 and pre- and immediately post- training session on day 2.
  Participants will rate on a scale of 0 (not confident at all) to 10 (extremely confident) their confidence in their ability to walk specified distances on the narrow beam.

SECONDARY OUTCOMES:
Change from baseline in average walking speed | Pre- and immediately post- training session on day 1 and pre- and immediately post- training session on day 2.
  Comfortable walking speed during traverses of 30ft laboratory
Change from baseline in narrow beam walking distance | Pre- and immediately post- training session on day 1 and pre- and immediately post- training session on day 2.
  Distance travelled on a low level narrow beam without stepping off
Change from baseline in horizontal ladder completion time | Pre- and immediately post- training session on day 1 and pre- and immediately post- training session on day 2.
  Time to traverse a horizontal ladder with randomly separated rungs.
Change from baseline in average step width during level walking | Pre- and immediately post- training session on day 1 and pre- and immediately post- training session on day 2.
  Mean width of right and left steps during traverses of 30ft laboratory
Change from baseline in average step length during level walking | Pre- and immediately post- training session on day 1 and pre- and immediately post- training session on day 2.
  Mean length of right and left steps during traverses of 30ft laboratory
Change from baseline in step width variability during level walking | Pre- and immediately post- training session on day 1 and pre- and immediately post- training session on day 2.
  Standard deviation of right and left step widths during traverses of 30ft laboratory

OTHER OUTCOMES:
Training protocol feasibility assessed by ability to complete 2-min bouts of walking on flat terrain | During training session on days 1 and 2 (each up to 45 minutes)
  Assessment of proposed duration of walking training bouts on flat terrain. For each of six training bouts, successful completion of 2-min of walking without trial termination will be recorded (yes/no).
Training protocol feasibility assessed by ability to complete 2-min bouts of walking on uneven terrain | During training session on days 1 and 2 (each up to 45 minutes)
  Assessment of proposed duration of walking training bouts on uneven terrain. For each of six training bouts, successful completion of 2-min of walking without trial termination will be recorded (yes/no).
Assessment protocol feasibility assessed by ability to take two steps or more on narrow beam | Immediately post- training sessions on days 1 and 2
  Assessment of feasibility of narrow beam-walking task. Ability to take at least two steps on a narrow beam after training session (yes/no).
Protocol acceptability assessed by session duration | During training session on days 1 and 2 (each up to 45 minutes)
  Duration of each session including testing and training in minutes.
Training protocol acceptability assessed by training acceptability questionnaire | Immediately after training on either day 1 or day 2
  Five item self-report Likert-style acceptability questionnaire, assessing the following components for uneven terrain training: 1) enjoyment, 2) challenge, 3) perceived safety, 4) tiredness after training, 5) desire to practice further

CONTACTS AND LOCATIONS:
Overall Officials: Jenny A Kent, PhD, Principal Investigator — University of Nevada, Las Vegas
Locations (1):
- University of Nevada Las Vegas, Las Vegas, Nevada, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Orsmond GI, Cohn ES. The Distinctive Features of a Feasibility Study: Objectives and Guiding Questions. OTJR (Thorofare N J). 2015 Jul;35(3):169-77. doi: 10.1177/1539449215578649. PMID 26594739
- [Background] Hanspal RS, Fisher K, Nieveen R. Prosthetic socket fit comfort score. Disabil Rehabil. 2003 Nov 18;25(22):1278-80. doi: 10.1080/09638280310001603983. PMID 14617445